CLINICAL TRIAL: NCT06743321
Title: A Prospective Study of the Effectiveness of Speech-to-speech Voice-cloning Care (SVCC) to Improve ICU-acquired Anxiety for Critically Ill Patients
Brief Title: Speech-to-speech Voice-cloning Care (SVCC) to Improve ICU-acquired Anxiety for Critically Ill Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K6842
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Critical Care Nursing
Keywords: ICU-acquired anxiety; Voice-cloning; Critical Care Nursing; Family-centered care; Artificial intelligence

STUDY DESIGN:
Masking Description: The independent statistician conducting the interim analysis will be masking. The statistician analyzing the primary and secondary outcome data will also be masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Patients in the intervention group will receive Speech-to-Speech Voice-Cloning Care (SVCC) as an addition to their standard ICU care.
  Interventions: Behavioral: Speech-to-speech Voice-Cloning Care (SVCC)
- The controlled group (No Intervention): Patients in the controlled group will only receive standard ICU care.

INTERVENTIONS:
Behavioral: Speech-to-speech Voice-Cloning Care (SVCC) — After patients in the intervention group were transferred to the ICU, the SVCC intervention was initiated. It is administered three times daily: in the morning, at noon, and in the evening. The SVCC intervention includes three types of activities: awakening, reassurance, and preparatory exercises for the removal of the endotracheal tube (ETT). Before each intervention is carried out, the clinical status of the participants must be assessed to determine whether they are suitable for SVCC and to decide on the specific content of the intervention. Once the removal of the ETT is implemented, the SVCC intervention will no longer be carried out.
  Arms: The intervention group

SUMMARY:
The goal of this clinical trial is to learn the effect of Speech-to-speech Voice-Cloning Care (SVCC) on improving ICU-acquired anxiety for critically ill patients. The main question it aims to answer is:

* Can the use of participants' loved ones' voices by nurses in communication while providing care lead to better mental health and clinical outcomes?

Researchers will see if the implementation of SVCC can reduce anxiety and depression and improve clinical outcomes.

Participants will:

* Receive the SVCC intervention until the endotracheal tube (ETT) is removed.
* Keep a diary of delirium, the duration of mechanical ventilation, and ICU stays.

DETAILED DESCRIPTION:
During the SVCC, healthcare will be delivered by nurses who will communicate with participants using the familiar voices of their loved ones, transformed in real-time by an artificial intelligence voice-cloning tool.

ELIGIBILITY:
Inclusion Criteria:

* Expected mechanical ventilation time > 24 hours;
* Expected ICU stay > 72 hours;
* Language: Chinese;
* Richmond Agitation-Sedation Scale (RAAS) score ≥ -2 points;
* Hemodynamic stability.

Exclusion Criteria:

* Severe hearing impairment or worse (Grade 3 or higher according to WHO's Grades of hearing impairment);
* Disorders of consciousness or comprehension;
* Mental or psychological disorders that are being treated with medication;
* Head trauma or surgery resulting in an inability to wear earphones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU-acquired anxiety | Baseline (Day 0); daily from ICU admission through ICU discharge (an average of 7 days); and 3 days post-ICU discharge.
  The primary outcome assessment will be conducted using the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A). The HADS is used to assess symptoms of anxiety and depression in medical patients, which includes two subscales: one for anxiety (HADS-A) and one for depression (HADS-D). Each subscale consists of seven items, with scores for each item ranging from 1 to 4. The total score for each subscale ranges from 7 to 28, with a score of 11 or above considered to be the critical value.

SECONDARY OUTCOMES:
ICU-acquired depression | Baseline (Day 0); daily from ICU admission through ICU discharge (an average of 7 days); and 3 days post-ICU discharge.
  ICU-acquired depression is assessed by the Hospital Anxiety and Depression Scale - Depression Subscale (HADS-D).
Incidence of Delirium | Twice daily from Day 1 through ICU discharge, an average of 7 days.
  The incidence of delirium is monitored and evaluated by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). The CAM-ICU has four items: (1) altered mental status/fluctuating course, (2)inattention, (3) altered level of consciousness, and (4) disorganized thinking. Each item has two factors (positive or negative). The physicians can diagnose the patients with delirium when the results of item (1), item (2), and item (3) or item (4) are positive.
Duration of Mechanical Ventilation | From the start of mechanical ventilation through endotracheal tube (ETT) removal, an average of 6 days.
  The duration of mechanical ventilation is daily recorded by the physicians and nurses.
ICU Stay | From ICU admission through ICU discharge, an average of 7 days.
  The ICU stays are daily recorded by the physicians and nurses.
Qualitative assessment | Once during the follow-up visit, three days after the participant is discharged from the ICU.
  To assess subjective patient experiences, brief, semi-structured interviews will be conducted with a subset of eligible participants in the intervention group to explore their perceptions, acceptance, and the impact of the voice-cloning intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Director — Peking union medical college hospital, ICU department
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not applicable due to the risk of patient privacy breaches and the potential for tampering with or leakage of patients' family members' voice data.

REFERENCES:
- [Background] Novaes MA, Knobel E, Karam CH, Andreoli PB, Laselva C. A simple intervention to improve satisfaction in patients and relatives. Intensive Care Med. 2001 May;27(5):937. doi: 10.1007/s001340100910. No abstract available. PMID 11430555
- [Background] Cray L. A collaborative project: initiating a family intervention program in a medical intensive care unit. Focus Crit Care. 1989 Jun;16(3):213-8. PMID 2737344
- [Background] May AD, Parker AM, Caldwell ES, Hough CL, Jutte JE, Gonzalez MS, Needham DM, Hosey MM. Provider-Documented Anxiety in the ICU: Prevalence, Risk Factors, and Associated Patient Outcomes. J Intensive Care Med. 2021 Dec;36(12):1424-1430. doi: 10.1177/0885066620956564. Epub 2020 Oct 9. PMID 33034254
- [Background] Fond G, Nemani K, Etchecopar-Etchart D, Loundou A, Goff DC, Lee SW, Lancon C, Auquier P, Baumstarck K, Llorca PM, Yon DK, Boyer L. Association Between Mental Health Disorders and Mortality Among Patients With COVID-19 in 7 Countries: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2021 Nov 1;78(11):1208-1217. doi: 10.1001/jamapsychiatry.2021.2274. PMID 34313711
- [Background] Rabiee A, Nikayin S, Hashem MD, Huang M, Dinglas VD, Bienvenu OJ, Turnbull AE, Needham DM. Depressive Symptoms After Critical Illness: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 Sep;44(9):1744-53. doi: 10.1097/CCM.0000000000001811. PMID 27153046
- [Background] Scragg P, Jones A, Fauvel N. Psychological problems following ICU treatment. Anaesthesia. 2001 Jan;56(1):9-14. doi: 10.1046/j.1365-2044.2001.01714.x. PMID 11167429
- [Background] Parker AM, Sricharoenchai T, Raparla S, Schneck KW, Bienvenu OJ, Needham DM. Posttraumatic stress disorder in critical illness survivors: a metaanalysis. Crit Care Med. 2015 May;43(5):1121-9. doi: 10.1097/CCM.0000000000000882. PMID 25654178
- [Background] Cuthbertson BH, Scott J, Strachan M, Kilonzo M, Vale L. Quality of life before and after intensive care. Anaesthesia. 2005 Apr;60(4):332-9. doi: 10.1111/j.1365-2044.2004.04109.x. PMID 15766335
- [Background] Jacques T, Ramnani A, Deshpande K, Kalfon P. Perceived Discomfort in Patients admitted to Intensive Care (DETECT DISCOMFORT 1): a prospective observational study. Crit Care Resusc. 2019 Jun;21(2):103-109. PMID 31142240
- [Background] Berntzen H, Bjork IT, Storsveen AM, Woien H. "Please mind the gap": A secondary analysis of discomfort and comfort in intensive care. J Clin Nurs. 2020 Jul;29(13-14):2441-2454. doi: 10.1111/jocn.15260. Epub 2020 Apr 17. PMID 32242994
- [Background] Baumgarten M, Poulsen I. Patients' experiences of being mechanically ventilated in an ICU: a qualitative metasynthesis. Scand J Caring Sci. 2015 Jun;29(2):205-14. doi: 10.1111/scs.12177. Epub 2014 Nov 7. PMID 25376648